CLINICAL TRIAL: NCT07183670
Title: Standardized Tracheostomy Decannulation Protocol for Patients With Prolonged Disorders of Consciousness: A Prospective Multicenter Cohort Study
Brief Title: Standardized Tracheostomy Decannulation Protocol for Patients With Prolonged Disorders of Consciousness
Acronym: STEP-DoC
Status: Not yet recruiting | Type: Observational
Sponsor: Hongying Jiang (Other)
Collaborators: Beijing Rehabilitation Hospital (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor-Investigator, Hongying Jiang, Principal Investigator, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: 2025-hxkfzx-step-doc
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Prolonged Disorders of Consciousness; Tracheostomy
Keywords: Decannulation; Protocol; Rehabilitation; Prolonged disorders of consciousness; Speaking wave

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Samples without DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decannulation Cohort: Patients who pass decannulation protocol
  Interventions: Diagnostic Test: decannulation protocol
- Not-decannulation Cohort: Patients failing at any protocol stage
  Interventions: Diagnostic Test: decannulation protocol

INTERVENTIONS:
Diagnostic Test: decannulation protocol — Step 1: The patient's clinical stability is confirmed. Step 2: Tolerance to the speaking valve is assessed. Step 3: The wearing time of the speaking valve is extended continuously for 4 h, and no tracheostomy cannula is used for sputum suction within 4 h.
  Step 4: Cough strength is evaluated to be good before decannulation. Decannulation Criteria: Pass Step 1 + Step 2 + Step 3 + Step 4

SUMMARY:
To evaluate the feasibility of a standardized tracheostomy decannulation protocol for patients with prolonged Disorders of Consciousness (pDoC) in rehabilitation hospitals.

DETAILED DESCRIPTION:
Advances in critical care have significantly increased the number of survivors with severe acquired brain injury (sABI). A subset of these patients develops Disorders of Consciousness (DoC), defined as prolonged DoC (pDoC) when lasting >28 days. Tracheostomy is often indicated for long-term mechanical ventilation and airway protection. However, tracheostomy tubes may cause inflammation, stenosis, excessive coughing, and dysphagia. Decannulation improves patient comfort, appearance, swallowing, communication, and social reintegration, while reducing long-term complications (e.g., tracheal stenosis, malacia, vocal cord injury, accidental decannulation) . Despite these benefits, consensus on safety and optimal timing for decannulation in pDoC remains elusive due to uncertain airway protection and aspiration risks. Our center previously demonstrated that a standardized decannulation protocol implemented by a pulmonary rehabilitation team correlates with successful decannulation. Key innovations include: (1) Replacing capping trials with 4-hour continuous tolerance of a speaking valve (reducing airway resistance and delayed decannulation ); (2) Not considering dysphagia a contraindication if patients manage secretions effectively and retain cough strength, even if requiring enteral nutrition (nasogastric/jejunal tubes or PEG) . This multicenter study aims to validate this protocol in pDoC patients and assess changes in consciousness levels pre-/post-decannulation.

ELIGIBILITY:
Inclusion Criteria:

1. CRS-R score >0
2. Signed informed consent by legal representative

Exclusion Criteria:

1. Non-PDOC tracheostomy patients
2. Death within 2 weeks post-referral
3. Active respiratory infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Condition: Prolonged Disorders of Consciousness (PDOC >28 days) Population: Tracheostomized adults in rehabilitation hospitals
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Decannulation rate | At decannulation protocol
  Proportion passing full protocol
Decannulation success rate | At 48 hours post decannulation
  (Decannulation - Decannulation failure ) / Decannulation

SECONDARY OUTCOMES:
CRS-R change rate | At a week post decannulation
  (Post-decannulation - Baseline)/Baseline
Time to decannulation | through study completion, an average of 1 year
  Days from referral to decannulation
Reintubation rate | 3-month follow-up
  Unplanned reintubation

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Jiang, Study Chair — Beijing Rehabilitation Hospital, Capital Medical University, Beijing
Locations (2):
- China (2):
  - Beijing Rehabilitation Hospital, Capital Medical University, Beijing,China, Beijing, Beijing Municipality
  - Beijing Rehabilitation Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hakiki B, Draghi F, Pancani S, Portaccio E, Grippo A, Binazzi B, Tofani A, Scarpino M, Macchi C, Cecchi F. Decannulation After a Severe Acquired Brain Injury. Arch Phys Med Rehabil. 2020 Nov;101(11):1906-1913. doi: 10.1016/j.apmr.2020.05.004. Epub 2020 May 16. PMID 32428445
- [Background] Draghi F, Pancani S, De Nisco A, Romoli AM, Maccanti D, Burali R, Grippo A, Macchi C, Cecchi F, Hakiki B. Implications of the Consciousness State on Decannulation in Patients With a Prolonged Disorder of Consciousness. Arch Phys Med Rehabil. 2024 Sep;105(9):1691-1699. doi: 10.1016/j.apmr.2024.05.006. Epub 2024 May 10. PMID 38734048
- [Background] Zhou T, Wang J, Zhang C, Zhang B, Guo H, Yang B, Li Q, Ge J, Li Y, Niu G, Gao H, Jiang H. Tracheostomy decannulation protocol in patients with prolonged tracheostomy referred to a rehabilitation hospital: a prospective cohort study. J Intensive Care. 2022 Jul 16;10(1):34. doi: 10.1186/s40560-022-00626-3. PMID 35842715